CLINICAL TRIAL: NCT06812117
Title: A Prospective, Observational, Multicenter Study to Evaluate the Safety and Effectiveness of Mirogabalin in Chinese Adult Patients With Diabetic Peripheral Neuropathic Pain (DPNP) in Real-world Clinical Practice Setting (ReMIssion Study)
Brief Title: A Study to Evaluate the Safety and Effectiveness of Mirogabalin in Chinese Adult Patients With Diabetic Peripheral Neuropathic Pain (DPNP) in Real-world Clinical Practice Setting (ReMIssion Study)
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS5565-0002-NIS-MA
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetic peripheral neuropathic pain; Real-world evidence; Mirogabalin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic peripheral neuropathic pain (DPNP): Patients diagnosed with DPNP and newly treated with mirogabalin.
  Interventions: Other: No Drug

INTERVENTIONS:
Other: No Drug — This is an non-interventional, observational study. No drug will be provided or administered as part of this protocol; however, participants on mirogabalin will be enrolled in this study.

SUMMARY:
This study will evaluate the safety and effectiveness of mirogabalin in adult patients with diabetic peripheral neuropathic pain (DPNP) in real-world clinical practice setting in China.

DETAILED DESCRIPTION:
Mirogabalin has been approved in China for the treatment of DPNP. Although there is evidence of the safety and efficacy of mirogabalin, there is a lack of real-world evidence on its safety and effectiveness to inform decision-making among a more diverse patient population in real-world clinical practice, such as patients with moderate or severe renal impairment; patients with more complications, comorbidities, and treatments; and patients with different severity of pain.

This study aims to collect safety and effectiveness data to guide physicians in the clinical use of mirogabalin for the treatment of patients with DPNP in the real-world clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be eligible for this study.

1. Age ≥ 18 years at the time of informed consent form (ICF) signed.
2. Patients diagnosed with DPNP (defined as patients diagnosed with type 1 or type 2 diabetes and painful distal symmetric polyneuropathy).
3. Patients with a pain scale of visual analog scale (VAS( ≥ 40 mm on the day of ICF signed.
4. Patients who are mirogabalin naïve prior to ICF signed and planned to initiate mirogabalin treatment.
5. Patients who are able to give signed ICF for study participation and willing to provide access to previous and future medical information.

Patients who meet any of the following criteria will be excluded from this study.

1. Patients who have other severe pain unrelated to DPN at baseline, which may confound the assessment of DPNP.
2. Patients who previously received pregabalin ≥ 300 mg/day or gabapentin ≥ 1200 mg/day to treat DPNP and declared lack of effectiveness.
3. Patients who received pregabalin, gabapentin, crisugabalin, or any other DPNP analgesic medications* within 7 days prior to ICF signed.

   *Other DPNP analgesic medication includes TCAs (amitriptyline, nortriptyline), SNRIs (duloxetine, venlafaxine), antiepileptics (carbamazepine), opioids (tapentadol, tramadol).
4. Patients with major psychiatric disorders (depression, Alzheimer disease, Parkinson disease, mania, bipolar disorder, psychosis, or schizophrenia, etc.) at baseline.
5. Patients with contraindications for mirogabalin treatment according to China package insert of mirogabalin.
6. Patients with simultaneous participation in any interventional clinical study.
7. Female patients at the status of pregnancy, potential pregnancy, or breast feeding.
8. Patients who have been judged by the investigator to be unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients diagnosed with DPNP and newly treated with mirogabalin will be consecutively enrolled in this study and followed up until the end of 15-week observation period, the end of 1-week observation period after the discontinuation of mirogabalin, withdrawal of consent, loss to follow-up, or study closure, whichever occurs first, to collect and evaluate patients' outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with any treatment related adverse events (TRAEs) | Baseline to Week 14
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Time-to-onset of somnolence, dizziness, weight gain, and peripheral edema | Baseline to Week 14
  For time-to-event variables, the median time, Q1 and Q3 as well as 95% CI will be estimated.
Symptom duration of somnolence, dizziness, weight gain, and peripheral edema | Baseline to Week 14
  For time-to-event variables, the median time, Q1 and Q3 as well as 95% CI will be estimated.
Proportion of participants with TEAEs, serious TEAEs, TRAEs leading to study treatment discontinuation | Baseline to Week 14
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Change from baseline in VAS pain | Week 14
  The VAS is used for the participant to rate average pain intensity of past 24 hours on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain. Reductions in VAS pain scores indicate better clinical outcome.
Proportion of participants achieving 30% and 50% pain relief (reduction in VAS score compared to baseline) | Baseline to Week 14
  The VAS is used for the participant to rate average pain intensity of past 24 hours on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain. Reductions in VAS pain scores indicate better clinical outcome.
Time to achieve 30% pain relief or 50% pain relief (reduction in VAS score compared to baseline) | Baseline to Week 14
  The VAS is used for the participant to rate average pain intensity of past 24 hours on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain. Reductions in VAS pain scores indicate better clinical outcome.
Change from baseline in Douleur Neuropathique 4 questions (DN4) score | Week 14
  DN4 will be assessed by the investigator after ICF signed and prior to the first administration of mirogabalin as baseline, when participants return to the clinical site during treatment period of mirogabalin, and at the end of mirogabalin treatment.
  Each "yes" answer is assigned 1 point, and a total score is calculated. A score of 4 or higher indicates a higher likelihood of neuropathic pain (eg. worse clinical outcome), while a score below 3 suggests it is less likely (eg. better clinical outcome).
Patient Global Impression of Change (PGIC) | Week 14
  Participants will provide a self-assessment using the 7-point scale via ePRO at the end of mirogabalin treatment: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse. Lower PGIC scores indicate better clinical outcome.
Change from baseline in EuroQol 5-Dimension 5-level (EQ-5D-5L) | Week 14
  The self-administered EQ-5D-5L includes the EQ-5D and the EQ VAS. EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3-moderate problems, 4=severe problems and 5=extreme problems. The patient is asked to indicate his/her health state in each of the five dimensions, resulting in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Lower 5-digit numbers indicates better clinical outcome (ie, health state).
  The EQ VAS records the patient's self-rated health on a vertical VAS where the endpoints are labelled '100 - The best health you can imagine' and '0 - The worst health you can imagine'. Higher EQ VAS scores indicate better clinical outcome/health.

CONTACTS AND LOCATIONS:
Overall Officials: Project Manager, Study Director — Daiichi Sankyo Co., Ltd.
Locations (30):
- China (30):
  - China-Japan friendship hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - Chengdu First People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First People's Hospital Of Foshan, Foshan
  - Shunde Hospital of southern Medical University, Foshan
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Affiliated Hospital of Henan University of Science & Technology, Henan
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - ZhongShan Hospital Fudan University, Shanghai
  - Shenzhen Nanshan People's Hospital, Shenzhen
  - First Hospital of Shanxi Medical University, Taiyuan
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Yibin Second People's Hospital, Yibin

IPD SHARING:
Plan to Share IPD: No